CLINICAL TRIAL: NCT02391480
Title: A Phase 1 Study Evaluating the Safety and Pharmacokinetics of ABBV-075 in Subjects With Advanced Cancer
Brief Title: A Study Evaluating the Safety and Pharmacokinetics of ABBV-075 in Subjects With Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M14-546
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2019-07

CONDITIONS: Cancer; Breast Cancer; Non-Small Cell Lung Cancer; Acute Myeloid Leukemia (AML); Multiple Myeloma; Prostate Cancer; Small Cell Lung Cancer; Non-Hodgkins Lymphoma
Keywords: Cancer; Bromodomain Inhibitor
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Leukemia, Myeloid, Acute; Multiple Myeloma; Prostatic Neoplasms; Small Cell Lung Carcinoma; Lymphoma, Non-Hodgkin | interventions — mivebresib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- ABBV-075 (Experimental): Dose escalation cohorts of ABBV-075 monotherapy
  Interventions: Drug: ABBV-075
- ABBV-075 and venetoclax combination (Experimental): Expansion cohorts of ABBV-075 and venetoclax combination therapy
  Interventions: Drug: ABBV-075; Drug: Venetoclax
- ABBV-075 expansion (Experimental): Expansion cohorts of ABBV-075 monotherapy
  Interventions: Drug: ABBV-075

INTERVENTIONS:
Drug: ABBV-075 — ABBV-075 Oral tablets
  Other Names: Mivebresib
Drug: Venetoclax — Venetoclax tablets, film-coated
  Other Names: Venclexta
  Arms: ABBV-075 and venetoclax combination

SUMMARY:
This is a Phase 1, first-in-human, dose escalation study in participants with advanced solid tumors to determine the pharmacokinetics, maximum tolerated dose and the recommended Phase 2 dose of ABBV-075 at different monotherapy dosing schedules. In addition the study will evaluate the safety. tolerability and the pharmacokinetics of ABBV-075 monotherapy or combination therapy in disease specific expansion cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Participant in the dose escalation cohorts must have histological confirmation of locally advanced or metastatic solid tumor that is either refractory after standard of care therapy for the disease or for which standard of care therapy or does not exist.
2. Participants in the expansion cohorts must have histological confirmation of AML, Multiple Myeloma, breast cancer, NSCLC, prostate cancer, SCLC, or NHL that is either refractory after standard of care therapy or for which standard of care therapy does not exist.
3. Participant must have an Eastern Cooperative Oncology Group (ECOG) Performance status of: 0 - 1 (dose escalation cohorts) or 0 - 2 (expansion cohorts)
4. Participants in the dose escalation cohort must have a serum albumin of ≥ 3.2 g/dL at screening.
5. Adequate bone marrow, renal, and hepatic function.
6. QTc interval < 480 milliseconds (msec) on the baseline electrocardiogram.

Exclusion Criteria:

1. Participant has untreated brain or meningeal metastases.
2. Participant has received anti-cancer therapy including chemotherapy, immunotherapy, biologic or any investigational therapy within a period of 21 days prior to Study Day 1.
3. Participant has active peptic ulcer disease or other hemorrhagic esophagitis/gastritis.
4. Symptoms of gross hematuria or gross hemoptysis.
5. Exhibits symptomatic or persistent, uncontrolled hypertension (BP > or = to 140 and/or diastolic pressure of > or = to 90 mm Hg).
6. History of long QT syndrome.
7. Peripheral neuropathy greater than or equal to grade 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2015-04-14 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-07-05 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of ABBV-075 | Minimum first cycle of dosing (28 days) up to one year for dose escalation segment.
  Maximum tolerated dose is defined as the highest dose level at which less than 2 of 6 participants experience the same dose limiting toxicity. If more than 2 participants experience a different dose limiting toxicity, the maximum tolerated dose may be further evaluated or determined to be exceeded based on discussions with the investigators and medical monitors.
Time to Cmax (peak time, Tmax) for ABBV-075 | Approximately 24 hours following a single dose of ABBV-075 up to approximately 2 years.
Number of participants with adverse events | Screening, Cycle 1 Day 1, 8 and 15, then Day 1 of each cycle up to approximately 2 years.
Maximum observed plasma concentration (Cmax) of ABBV-075 | Approximately 24 hours following a single dose of ABBV-075 up to approximately 2 years.
Area under the curve (AUC) | Cycle 1 Day 1 Pre-dose, 1, 2, 3, 4, 6, 8 and 24 hours post ABBV-075 dosing, and on Cycle 1 Day 15 at 14, 17, 20 hours post dose.
  Area under the plasma concentration versus time curve from time 0 (pre-dose) to the time of the last measurable concentration (AUC 0-t).

SECONDARY OUTCOMES:
Duration of overall response (DOR) | At screening, every 8 weeks from Cycle 1 Day 1, and at the Final visit up to approximately 2 years.
  DOR is defined as the time from the participant's initial CR or PR to the time of disease progression
Objective Response Rate (ORR) | At screening, every 8 weeks from Cycle 1 Day 1, and at the Final visit up to approximately 2 years.
  ORR is defined as the proportion of participants who have a complete response (CR) or partial response (PR).
Progression Free Survival (PFS) | Screening, every 8 weeks from Cycle 1 Day 1, and at the Final visit up to approximately 2 years.
  PFS is defined as the time from the first dose of ABBV-075 to either disease progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (10):
- United States (10):
  - Scottsdale Healthcare /ID# 132963, Scottsdale, Arizona
  - City of Hope /ID# 154053, Duarte, California
  - UC Davis Comp Cancer Ctr /ID# 154644, Sacramento, California
  - Yale University /ID# 136982, New Haven, Connecticut
  - University of Chicago /ID# 155453, Chicago, Illinois
  - Indiana Univ School Medicine /ID# 132946, Indianapolis, Indiana
  - Duke Univ Med Ctr /ID# 154647, Durham, North Carolina
  - Mary Crowley Cancer Research /ID# 154059, Dallas, Texas
  - Univ TX, MD Anderson /ID# 132276, Houston, Texas
  - UT MD Anderson Cancer Center /ID# 164122, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Piha-Paul SA, Sachdev JC, Barve M, LoRusso P, Szmulewitz R, Patel SP, Lara PN Jr, Chen X, Hu B, Freise KJ, Modi D, Sood A, Hutti JE, Wolff J, O'Neil BH. First-in-Human Study of Mivebresib (ABBV-075), an Oral Pan-Inhibitor of Bromodomain and Extra Terminal Proteins, in Patients with Relapsed/Refractory Solid Tumors. Clin Cancer Res. 2019 Nov 1;25(21):6309-6319. doi: 10.1158/1078-0432.CCR-19-0578. Epub 2019 Aug 16. PMID 31420359
- [Derived] Borthakur G, Odenike O, Aldoss I, Rizzieri DA, Prebet T, Chen C, Popovic R, Modi DA, Joshi RH, Wolff JE, Jonas BA. A phase 1 study of the pan-bromodomain and extraterminal inhibitor mivebresib (ABBV-075) alone or in combination with venetoclax in patients with relapsed/refractory acute myeloid leukemia. Cancer. 2021 Aug 15;127(16):2943-2953. doi: 10.1002/cncr.33590. Epub 2021 May 2. PMID 33934351